CLINICAL TRIAL: NCT01384968
Title: Acute Dietary Nitrate Supplementation to Improve Performance in Endurance Trained Athletes
Brief Title: Acute Nitrate Supplementation in Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 11-3-033
Record Dates: First submitted 2011-06-23; First posted 2011-06-29 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Acute Nitrate Ingestion on Athletic Performance
Keywords: nitrite; exercise; cycling
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beetroot juice (Experimental): beetroot juice (170 mL, 8 mmol nitrate)
  Interventions: Dietary Supplement: beetroot juice
- Nitrate-depleted beetroot juice (Placebo Comparator): 140 mL ...0 nitrate. Beetroot juice
  Interventions: Dietary Supplement: beetroot juice

INTERVENTIONS:
Dietary Supplement: beetroot juice — 170 mL beetroot juice (Beet It, James White drinks Ltd).
  Other Names: Beet It, James White Drinks Ltd.

SUMMARY:
Six days of dietary nitrate (NO3-) supplementation in the form of beetroot juice (~0.5 L•d-1; 5.1-11.2 mmol NO3- •d-1) has been purported to reduce pulmonary oxygen uptake (VO2) during submaximal exercise and increase tolerance to high-intensity workloads. These results suggest that dietary nitrate supplementation has the potential to act as an ergogenic aid. Recently, we assessed submaximal oxygen uptake and 10 km time trial performance after 6 d of dietary nitrate supplementation in trained cyclists. We demonstrated an improvement in time trial performance compared to the nitrate-depleted placebo. However, the minimal dosage and duration of nitrate supplementation that is needed to elicit these performance effects remain largely unknown. Therefore, the purpose of the study is to assess performance capacity following an acute dose of nitrate supplementation consumed 3 h prior to the onset of exercise in trained cyclists. We will test the hypothesis that a single dose (140 mL; ~8 mmol NO3-) of dietary nitrate supplementation in the form of beetroot juice, ingested 3 h prior to exercise will improve time trial performance in trained cyclists compared to a nitrate-depleted placebo.

DETAILED DESCRIPTION:
Recent work in humans suggests that increasing nitric oxide (NO) bioavailability may induce physiological changes beyond the well known hemodynamic effects (Dejam, Hunter et al. 2004; Webb, Patel et al. 2008). NO plays a key role in the regulation of blood flow, muscle contractility, myocyte differentiation, glucose and calcium homeostasis (Dejam, Hunter et al. 2004). Within the human body, exogenous nitrate (NO3-) which has a half-life of 6-7 hours (h) (Lundberg, Weitzberg et al. 2008) is reduced to bioactive nitrite (NO2-) by facultative anaerobic bacteria in the saliva and further to NO via various pathways (Duncan, Dougall et al. 1995; Zhang, Naughton et al. 1998). Several groups (Larsen, Weitzberg et al. 2007; Bailey, Fulford et al. 2009; Bailey, Winyard et al. 2010; Larsen, Weitzberg et al. 2010; Vanhatalo, Bailey et al. 2010; Lansley, Winyard et al. 2011) have investigated whether dietary nitrate provision affects metabolic or circulatory parameters during exercise in vivo in humans. Oral ingestion of sodium nitrate (0.1 mmol•kg-1•d-1) for 2-3 days (d) has been shown to significantly reduce pulmonary oxygen uptake (VO2) during submaximal cycling exercise in both untrained (Larsen, Weitzberg et al. 2010) and trained men (Larsen, Weitzberg et al. 2007). Since the use of sodium nitrate is regulated in most countries, researchers have started to examine the impact of ingesting nitrate-rich foods, such as beetroot juice, on the physiological response to exercise (Bailey, Fulford et al. 2009; Bailey, Winyard et al. 2010; Vanhatalo, Bailey et al. 2010; Lansley, Winyard et al. 2011).

Recent work by Jones and colleagues have demonstrated that ingestion of 0.5 L beetroot juice per d for 6 d reduces pulmonary oxygen uptake during submaximal exercise (Bailey, Fulford et al. 2009; Vanhatalo, Bailey et al. 2010; Lansley, Winyard et al. 2011) and lowers the ATP cost of muscle force production suggesting an enhanced contractile efficiency (Bailey, Winyard et al. 2010). This improvement in exercise efficiency was evident acutely (2.5 h) after ingestion of a single 0.5 L bolus of beetroot and persisted for 15 d when supplementation was continued (Vanhatalo, Bailey et al. 2010). Although the active ingredient in beetroot has been assumed to be nitrate, beetroot is rich in several other potentially metabolically-active compounds (e.g. polyphenols). To confirm whether the proposed cardiovascular and physiological benefits of beetroot juice are solely attributable to its high NO3- content, Jones and colleagues tested beetroot juice against nitrate-depleted beetroot juice. They verified their previous findings (Bailey, Fulford et al. 2009) by demonstrating a lowered O2 cost of submaximal exercise following ingestion of 0.5 L beetroot juice for 6 d when compared with the nitrate-depleted juice (Lansley, Winyard et al. 2011).

From the proposed improvements in metabolic efficiency, it has been suggested that nitrate supplementation (0.5 L•d-1; ~5.1-11.2 mmol NO3- •d-1) may increase exercise tolerance or time to fatigue when exercise is performed at higher workloads (Bailey, Fulford et al. 2009; Bailey, Winyard et al. 2010; Vanhatalo, Bailey et al. 2010; Lansley, Winyard et al. 2011). The latter suggests that inorganic nitrate ingestion may act as a strong ergogenic aid. We recently tested the potential ergogenic properties of nitrate using a more practical, performance-based study that simulated athletic competition in a trained subject population (Cermak, Gibala et al. 2011). We demonstrated that following 6 d of dietary nitrate supplementation in the form of concentrated beetroot juice (140 mL•d-1; ~4 mmol NO3- •d-1), mean VO2 was lower during submaximal exercise and 10 km time-trial performance improved in trained cyclists (Cermak, Gibala et al. 2011). However, the minimal dosage and duration of nitrate supplementation that is needed to elicit these performance effects remains largely unknown. Although time to exhaustion is not a very practical performance measurement, improvements in such performance tests have been observed after only 4 d of dietary nitrate supplementation (0.5 L•d-1; ~6.2 mmol•d-1 NO3-). Furthermore, even a single dose of nitrate (~5.2 mmol NO3-) has been shown to lower mean VO2 values measured 2.5 h after ingesting 0.5 L of beetroot juice (Vanhatalo, Bailey et al. 2010). Whether a similar improvement in time-trial performance would also be observed after a shorter supplementation period is presently unknown. Therefore, the present study aims to investigate whether a single dose of dietary nitrate (140 mL; ~8 mmol NO3-) ingested 3 h prior to the onset of exercise will improve time-trial performance in trained cyclists.

Furthermore, inorganic nitrate ingestion (beetroot juice) has also been demonstrated to improve time to claudication pain while walking in peripheral artery disease patients (Kenjale, Ham et al. 2011), and lower plasma triglycerides in patients at risk for cardiovascular disease (Zand, Lanza et al. 2011), providing evidence for inorganic nitrate ingestion to improve vasodilation/perfusion. Whether a bolus ingestion of nitrate would also influence the perfusion of nutrients following the ingestion of a small meal remains unknown. Therefore, in a secondary aim, we want to investigate the plasma metabolite response in addition to nitrate and nitrite concentrations following the nitrate supplementation and subsequent meal ingestion.

1. OBJECTIVES The main objective will be to identify whether a bolus (140 mL) ingestion of dietary nitrate (~8 mmol NO3-) in the form of concentrated beetroot juice will acutely increase time-trial performance compared to a nitrate-depleted placebo (140 mL; ~0.0047 mmol NO3-). A secondary objective will be to measure blood samples after nitrate and meal ingestion to assess any changes in the concentration of nitrate, nitrite, glucose, insulin, lactate and free fatty acids. In this secondary objective, we are most interested in determining whether nitrate supplementation changes blood metabolites (glucose, insulin, lactate, free fatty acids) following 1) meal ingestion and 2) immediate post-exercise recovery period in comparison to the placebo. We will test the hypothesis that a single dose (140 mL; ~8 mmol NO3-) of dietary nitrate supplementation (beetroot juice) ingested 3 h prior to exercise will improve time-trial performance in trained cyclists compared to the nitrate-depleted placebo.
2. STUDY DESIGN (Protocol) After the assessment of aerobic capacity (step-wise exercise cycling test to exhaustion) and familiarization testing, subjects will be randomized in a double-blind fashion to the treatment order of a bolus ingestion of nitrate (beetroot juice) and placebo (nitrate-depleted beetroot juice). For the two experimental trials, subjects will report to the laboratory at 8.00 h for the insertion of the blood catheter into an antecubital vein. Subjects will then be asked to consume 140 mL of either concentrated beetroot juice nitrate or concentrated nitrate-depleted beetroot juice (placebo). Following the consumption of the beverage, subjects will be given a standardized breakfast and will then rest in the lab for 2.5 h before being weighed and fitted with a heart-rate monitor for the commencement of the time-trial (3 h post ingestion of treatment beverage). Blood samples will be drawn at time 0 min (before beverage ingestion), 30, 60, 90, 120, 150, 180 min (start of time-trial). Two more blood samples will be drawn immediately post and 30 minutes post time-trial (Figure 1). Sampling will occur every 30 minutes based on previous research examining blood metabolites following meal ingestion or an oral glucose load (van Dijk, Manders et al. 2011) and nitrate/nitrite concentrations (Webb, Patel et al. 2008). The last two blood samples will occur immediately following the time-trial and 30 min into the recovery period to assess any changes in metabolites and nitrate/nitrite concentrations from the exercise and during the short-term recovery period.

To assess time-trial performance, subjects will be instructed to perform a set amount of work in the shortest time possible. Total work to be performed will be calculated according to the equation of Jeukendrup, Saris, Brouns, and Kester (Jeukendrup, Saris et al. 1996), adapted by our lab (Beelen, Berghuis et al. 2009) :

Total amount of work = 0.60 • Wmax • 3,600

where Wmax is the maximal workload capacity determined during Visit 1 and 3,600 is the duration in seconds (equivalent to 1 hr). The ergometer will be set in linear mode to obtain 60% Wmax when subjects' cycle at their preferred cadence determined during Visit 1. The ergometer will be connected to a computer that will calculate and display the total amount of work performed. Subjects will receive no verbal or physiological feedback during the time-trial. The only information subjects will receive is the absolute amount of work performed and the percentage of total work performed relative to the set amount of work that needs to be completed. A fan will be placed 1 meter behind each participant to provide cooling and air circulation during the trials. Heart rate (Polar, Finland) will be recorded continuously throughout the test. This type of time-trial has been validated and used before in our lab (Beelen, Berghuis et al. 2009), for an overview of validation studies see (Currell and Jeukendrup 2008). Examples of coefficients of variation in similar trials are 1.1 (Palmer, Dennis et al. 1996), 0.7 (Smith, Davison et al. 2001) and 0.9 (Laursen, Shing et al. 2003). Water will be provided ad libitum during visits 1 and 2. However, the water consumed during visit 2 (familiarization trial) will be measured and repeated for visits 3 and 4 (exercise trials).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* 18 - 30 years of age
* Endurance cycling trained (≥3 sessions of endurance exercise per week)
* VO2 max ≥ 50 ml/kg/min
* Training history of more than one year of ≥3 sessions of endurance cycling exercise per week
* BMI <25 kg/m2

Exclusion Criteria:

* Use of medication
* Smoking
* Currently supplementing diet with beetroot juice

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Time-trial performance | Laboratory visits 2, 3 and 4 (each visit separated by ~ 1wk))
  Subjects will be asked to visit the laboratory for a total of 4 visits over 4 weeks. During visits 2,3 and 4 time-trial performance will be assessed. Each visit will be separated on average by at least 1 week. Therefore, if subjects have their first visit (max text) in week 1, their time trial performance will be assessed during weeks 2, 3 and 4.

SECONDARY OUTCOMES:
Nitrate and nitrite plasma concentration | Laboratory visits 3 and 4 (approximately 1 wk apart)
  During visits 3 and 4 (during the 4 week study), subjects will undergo blood sampling whereby we will assess plasma concentration for nitrate and nitrite. Each visit will be separated by approximately 1 week. Therefore, if subjects enroll in the study during week 1, we will assess nitrate and nitrite during weeks 3 and 4.
blood metabolites (glucose, insulin, lactate, free fatty acids) | Laboratory visits 3 and 4 (approximately 1 wk apart)
  During visits 3 and 4, subjects will undergo blood sampling whereby we will assess plasma concentration for blood metabolites (glucose, insulin, lactate and free fatty acids). Each visit will be separated by approximately 1 week. Therefore, if subjects enroll in the study during week 1, we will assess blood metabolites during weeks 3 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, Ph.D., Study Director — Maastricht University; Naomi Cermak, Ph.D., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Vanhatalo A, Bailey SJ, Blackwell JR, DiMenna FJ, Pavey TG, Wilkerson DP, Benjamin N, Winyard PG, Jones AM. Acute and chronic effects of dietary nitrate supplementation on blood pressure and the physiological responses to moderate-intensity and incremental exercise. Am J Physiol Regul Integr Comp Physiol. 2010 Oct;299(4):R1121-31. doi: 10.1152/ajpregu.00206.2010. Epub 2010 Aug 11. PMID 20702806
- [Background] Bailey SJ, Winyard P, Vanhatalo A, Blackwell JR, Dimenna FJ, Wilkerson DP, Tarr J, Benjamin N, Jones AM. Dietary nitrate supplementation reduces the O2 cost of low-intensity exercise and enhances tolerance to high-intensity exercise in humans. J Appl Physiol (1985). 2009 Oct;107(4):1144-55. doi: 10.1152/japplphysiol.00722.2009. Epub 2009 Aug 6. PMID 19661447
- [Background] Lansley KE, Winyard PG, Fulford J, Vanhatalo A, Bailey SJ, Blackwell JR, DiMenna FJ, Gilchrist M, Benjamin N, Jones AM. Dietary nitrate supplementation reduces the O2 cost of walking and running: a placebo-controlled study. J Appl Physiol (1985). 2011 Mar;110(3):591-600. doi: 10.1152/japplphysiol.01070.2010. Epub 2010 Nov 11. PMID 21071588
- [Background] Kenjale AA, Ham KL, Stabler T, Robbins JL, Johnson JL, Vanbruggen M, Privette G, Yim E, Kraus WE, Allen JD. Dietary nitrate supplementation enhances exercise performance in peripheral arterial disease. J Appl Physiol (1985). 2011 Jun;110(6):1582-91. doi: 10.1152/japplphysiol.00071.2011. Epub 2011 Mar 31. PMID 21454745
- [Background] Bailey SJ, Fulford J, Vanhatalo A, Winyard PG, Blackwell JR, DiMenna FJ, Wilkerson DP, Benjamin N, Jones AM. Dietary nitrate supplementation enhances muscle contractile efficiency during knee-extensor exercise in humans. J Appl Physiol (1985). 2010 Jul;109(1):135-48. doi: 10.1152/japplphysiol.00046.2010. Epub 2010 May 13. PMID 20466802
- [Background] Beelen M, Berghuis J, Bonaparte B, Ballak SB, Jeukendrup AE, van Loon LJ. Carbohydrate mouth rinsing in the fed state: lack of enhancement of time-trial performance. Int J Sport Nutr Exerc Metab. 2009 Aug;19(4):400-9. doi: 10.1123/ijsnem.19.4.400. PMID 19827464
- [Background] Cermak NM, Gibala MJ, van Loon LJ. Nitrate supplementation's improvement of 10-km time-trial performance in trained cyclists. Int J Sport Nutr Exerc Metab. 2012 Feb;22(1):64-71. doi: 10.1123/ijsnem.22.1.64. PMID 22248502
- [Background] Currell K, Jeukendrup AE. Validity, reliability and sensitivity of measures of sporting performance. Sports Med. 2008;38(4):297-316. doi: 10.2165/00007256-200838040-00003. PMID 18348590
- [Background] Dejam A, Hunter CJ, Schechter AN, Gladwin MT. Emerging role of nitrite in human biology. Blood Cells Mol Dis. 2004 May-Jun;32(3):423-9. doi: 10.1016/j.bcmd.2004.02.002. PMID 15121102
- [Background] Duncan C, Dougall H, Johnston P, Green S, Brogan R, Leifert C, Smith L, Golden M, Benjamin N. Chemical generation of nitric oxide in the mouth from the enterosalivary circulation of dietary nitrate. Nat Med. 1995 Jun;1(6):546-51. doi: 10.1038/nm0695-546. PMID 7585121
- [Background] Jeukendrup A, Saris WH, Brouns F, Kester AD. A new validated endurance performance test. Med Sci Sports Exerc. 1996 Feb;28(2):266-70. doi: 10.1097/00005768-199602000-00017. PMID 8775164
- [Background] Larsen FJ, Weitzberg E, Lundberg JO, Ekblom B. Effects of dietary nitrate on oxygen cost during exercise. Acta Physiol (Oxf). 2007 Sep;191(1):59-66. doi: 10.1111/j.1748-1716.2007.01713.x. Epub 2007 Jul 17. PMID 17635415
- [Background] Larsen FJ, Weitzberg E, Lundberg JO, Ekblom B. Dietary nitrate reduces maximal oxygen consumption while maintaining work performance in maximal exercise. Free Radic Biol Med. 2010 Jan 15;48(2):342-7. doi: 10.1016/j.freeradbiomed.2009.11.006. Epub 2009 Nov 12. PMID 19913611
- [Background] Laursen PB, Shing CM, Jenkins DG. Reproducibility of a laboratory-based 40-km cycle time-trial on a stationary wind-trainer in highly trained cyclists. Int J Sports Med. 2003 Oct;24(7):481-5. doi: 10.1055/s-2003-42012. PMID 12968204
- [Background] Lundberg JO, Weitzberg E, Gladwin MT. The nitrate-nitrite-nitric oxide pathway in physiology and therapeutics. Nat Rev Drug Discov. 2008 Feb;7(2):156-67. doi: 10.1038/nrd2466. PMID 18167491
- [Background] Palmer GS, Dennis SC, Noakes TD, Hawley JA. Assessment of the reproducibility of performance testing on an air-braked cycle ergometer. Int J Sports Med. 1996 May;17(4):293-8. doi: 10.1055/s-2007-972849. PMID 8814512
- [Background] Smith MF, Davison RC, Balmer J, Bird SR. Reliability of mean power recorded during indoor and outdoor self-paced 40 km cycling time-trials. Int J Sports Med. 2001 May;22(4):270-4. doi: 10.1055/s-2001-13813. PMID 11414669
- [Background] van Dijk JW, Manders RJ, Hartgens F, Stehouwer CD, Praet SF, van Loon LJ. Postprandial hyperglycemia is highly prevalent throughout the day in type 2 diabetes patients. Diabetes Res Clin Pract. 2011 Jul;93(1):31-7. doi: 10.1016/j.diabres.2011.03.021. Epub 2011 Apr 16. PMID 21497935
- [Background] Webb AJ, Patel N, Loukogeorgakis S, Okorie M, Aboud Z, Misra S, Rashid R, Miall P, Deanfield J, Benjamin N, MacAllister R, Hobbs AJ, Ahluwalia A. Acute blood pressure lowering, vasoprotective, and antiplatelet properties of dietary nitrate via bioconversion to nitrite. Hypertension. 2008 Mar;51(3):784-90. doi: 10.1161/HYPERTENSIONAHA.107.103523. Epub 2008 Feb 4. PMID 18250365
- [Background] Zand J, Lanza F, Garg HK, Bryan NS. All-natural nitrite and nitrate containing dietary supplement promotes nitric oxide production and reduces triglycerides in humans. Nutr Res. 2011 Apr;31(4):262-9. doi: 10.1016/j.nutres.2011.03.008. PMID 21530799
- [Background] Zhang Z, Naughton D, Winyard PG, Benjamin N, Blake DR, Symons MC. Generation of nitric oxide by a nitrite reductase activity of xanthine oxidase: a potential pathway for nitric oxide formation in the absence of nitric oxide synthase activity. Biochem Biophys Res Commun. 1998 Aug 28;249(3):767-72. doi: 10.1006/bbrc.1998.9226. PMID 9731211